CLINICAL TRIAL: NCT01862237
Title: Does Type II Diabetes Influence Prognosis and Left Ventricular Remodeling in Patients With Aortic Valve Stenosis Referred for Aortic Valve Replacement ?
Brief Title: Type II Diabetes Influence on Left Ventricular Remodeling and Outcomes in Patients Undergoing Aortic Valve Replacement Surgery.
Acronym: DIAPASON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011.699
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Type II Diabetes
Keywords: Type II diabetes; aortic valve stenosis; left ventricular remodeling; aortic valve replacement surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Aortic Valve Stenosis; Ventricular Remodeling | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with type II diabetes (Experimental): Type II diabetes patients with aortic valve stenosis referred for aortic valve replacement.
  Interventions: Other: Intervention
- Patients without type II diabetes (Experimental): No type II diabetes patients with aortic valve stenosis referred for aortic valve replacement.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — * blood collection
  * Completion of a pre-operative cardiac MRI.
  * Completion of a coronary angiography examination
  * Completion during the surgery d'une myocardial biopsy,
  * Aortic echocardiographic follow-up (including post-operative ultrasound and ultrasound at 1 year
  * Completion of a cardiac MRI 1 year after surgery.

SUMMARY:
This project focuses on the physiopathology of left ventricular remodeling associated with type II diabetes in patients with aortic valve stenosis referred for surgical aortic valve replacement.

The main objective is to compare the reverse left ventricular remodeling between patients with type II diabetes and case-control patients without diabetes at one(1) year after surgical aortic valve replacement.

The secondary objectives are :

1. assess the influence of type II diabetes on left ventricular remodeling in patients presenting with aortic valve stenosis,
2. assess the predictive value of myocardial fibrosis and other LV characteristics present prior to aortic valve surgery on the LV reverse remodeling and their influence on cardiovascular events at one (1) year after surgery,
3. assess the influence of type II diabetes on cardiovascular morbidity and mortality post aortic valve surgery.

The investigators main hypothesis is that patients with type II diabetes and aortic valve stenosis requiring aortic valve replacement have poorer LV function and less favorable post surgery clinical outcomes than patients without type II diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Arm 1: Treated Type II diabetes, Arm 2: absence of type II diabetes
* Aortic valve stenosis
* LVEF > 50% with no kinetic abnormalities
* Non significant obstructive coronary artery disease
* Absence of gadolinium enhanced MRI contraindications
* Informed consent signed
* Patient affiliated to the French Social Security.

Exclusion Criteria:

* Chronic arrhythmia or absence of sinus rhythm
* Past history of cardiomyopathy or coronary insufficiency
* Significant coronaropathy seen during the coronary angiography with >50% degree stenosis prior to aortic valve replacement
* Hemodynamically significant valvular dysfunction other than aortic stenosis (grade 2 mitral or aortic insufficiency, mitral valve stenosis < 1.5 cm2)
* Systemic chronic inflammatory disease leading to cardiac injury (scleroderma)
* Renal insufficiency (clearance < 30 ml/min)
* Insufficient transthoracic echocardiography echogenicity
* Type I diabetes mellitus
* Uncontrolled hypertension (> 180/100 mm Hg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Mass measured by echocardiography | Primary outcome is assessed at one year 1 year after aortic valve replacement.

SECONDARY OUTCOMES:
cardiovascular events (cardiac mortality, heart failure, atrial or ventricular rhythm abnormalities) and clinical improvement (NYHA class, 6-minute walk test). | 1 year after aortic valve replacement.
Measurement of BNP (Brain Natriuretic Peptide). | 1 year after aortic valve replacement.
Echocardiographic parameters. | 1 year after aortic valve replacement.
  Left Ventricular Ejection Fraction, Systolic Longitudinal Strain, Systolic Circumferential Strain, Systolic Radial Strain, Diameters, wall thickness.
Magnetic Resonance Imaging (MRI) parameters. | 1 year after aortic valve replacement.
  LV mass, volumes, ejection fraction, replacement fibrosis mass on delayed enhanced studies, and interstitial fibrosis quantification (T1 mapping studies).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Louis Pradel, Lyon, France

REFERENCES:
- [Derived] Cherpaz M, Meugnier E, Seillier G, Pozzi M, Pierrard R, Leboube S, Farhat F, Vola M, Obadia JF, Amaz C, Chalabreysse L, May C, Chanon S, Brun C, Givre L, Bidaux G, Mewton N, Derumeaux G, Bergerot C, Paillard M, Thibault H. Myocardial transcriptomic analysis of diabetic patients with aortic stenosis: key role for mitochondrial calcium signaling. Cardiovasc Diabetol. 2024 Jul 8;23(1):239. doi: 10.1186/s12933-024-02329-5. PMID 38978010